CLINICAL TRIAL: NCT01672502
Title: Fire Fighter Fatigue Management Program: Operation Fight Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Federal Emergency Management Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Charles Andrew Czeisler, MD, PhD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMW-2010-FP-00521
Record Dates: First submitted 2012-08-16; First posted 2012-08-27 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Shift-Work Sleep Disorder; Insomnia; Restless Leg Syndrome; Obstructive Sleep Apnea; Impaired Driving
Keywords: sleep; firefighter; fire; apnea; insomnia; shift; narcolepsy; restless leg; rls; fatigue; Optalert; actigraph; actigraphy; actiwatch; safety; sleepiness; sleepy; work; hours; FEMA; drowsy
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Restless Legs Syndrome; Sleep Apnea, Obstructive; Apnea; Narcolepsy; Fatigue; Sleepiness | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Firefighters in this group will receive at the beginning of the study an introduction to the study, sleep education, sleep disorder screening survey, health survey, increased sleep opportunities at their fire department, followed later by physiological monitoring of a portion of the firefighters, and then finally an 'end of year' survey at the end of the study.
  Interventions: Behavioral: Sleep health education provided via a web-based program; Other: Sleep disorder detection and treatment; Other: Optimization of Sleep in Fire Station
- Control (Active Comparator): Firefighters in this group will only receive an introduction to the study and a health survey, followed later by physiological monitoring of a portion of the firefighters, and then at the end of the study will receive the sleep disorders screening survey, sleep education (Intervention group received screening survey and education much earlier at the beginning of the study), and an 'end of year' survey. None of these firefighters will receive the increased sleep opportunities as the Intervention group will.
  Interventions: Behavioral: Sleep health education provided via a web-based program; Other: Sleep disorder detection and treatment

INTERVENTIONS:
Behavioral: Sleep health education provided via a web-based program — All firefighters in the experimental group and controls will be asked to complete an approximately 30 minute education session. This education session will split into two modules, module 1: an introduction to the program along with basic sleeps hygiene information and module 2: standard training. Topics covered in module 2 will include basic sleep physiology, the causes and consequences of sleep disorders, and fatigue countermeasures. We will emphasize strategies to maximize sleep and reduce fatigue both on and off work.
  Other Names: Operation Fight Fatigue; OFF; Comprehensive Fatigue Management Training Program
Other: Sleep disorder detection and treatment — Firefighters in the intervention districts will complete a sleep disorders screening questionnaire. The questionnaire will focus on identifying individuals who show increased likelihood of suffering from obstructive sleep apnea, insomnia, shift work disorder, and restless legs syndrome using validated screening tools. Those assessed to be at high risk for one of these sleep disorders will be referred to a local AASM-accredited Clinical Sleep Disorders Service for evaluation and, if necessary, treatment. Diagnosis and treatment of sleep-related disorders will reduce the risk of fatigue-related accidents and improve the health and safety of affected individuals.
  Other Names: Operation Fight Fatigue; OFF; Comprehensive Fatigue Management Training Program
Other: Optimization of Sleep in Fire Station — First, we will review and retrofit the sleeping quarters to provide a better environment for napping and sleep; light, noise, bed type, space, temperature, and location would all be considered and where possible, changes made to improve the sleeping environment. Secondly, we will work with management and union personnel to develop a 'sleep friendly' policy during the daytime, with specified protected times for naps during the day before the overnight work in order to reduce sleepiness during overnight work. Finally, we will upgrade the alerting systems, that is, we will work with management and union personnel to consider changing the policy that requires the sleeping areas of all stations to receive all alarm calls, even if that particular station is not required to attend the alarm.
  Other Names: Operation Fight Fatigue; OFF; Comprehensive Fatigue Management Training Program
  Arms: Intervention

SUMMARY:
Firefighters frequently work extended duration shifts and long work weeks which have adverse effects on alertness, health, safety and performance. This protocol uses a survey instrument to examine the effects of extended duration shifts on safety outcomes (e.g., motor vehicle crashes, accidents, injuries), health (e.g., diagnosis and treatment of sleep disorders, improved general health indices, decreased number of sick days), and performance (e.g., decreased response time). This study will expand understanding of the nature, scope, etiology and consequences of firefighter fatigue and increase our ability to develop guidelines that can be generalized across fire departments throughout North America. This study could provide an avenue to make lasting policy improvements that could enhance the safety, health, and performance of firefighters.

DETAILED DESCRIPTION:
Firefighters work some of the most challenging schedules known under highly stressful and demanding conditions. The need to work frequent extended shifts leads to acute and chronic sleep deficiency as well as disruption of circadian rhythms. Firefighters on-call overnight are also particularly susceptible to sleep inertia, the neurocognitive impairment experienced immediately upon waking. In addition, it is likely that a significant proportion of firefighters suffer from undiagnosed sleep disorders, which further impair sleep and exacerbate fatigue.

The proposed fatigue countermeasure aims to increase sleep opportunities, and thereby improve firefighter safety and health. We will be conducting a station-level, randomized clinical trial of policies designed to maximize sleep opportunities during current 24-hour shifts to improve alertness, performance, health and safety in firefighters.

We will leverage the comprehensive fatigue management program we developed and the web-based technology we implemented in previous Federal Emergency Management Agency projects, and will continue to offer our web-based education program and sleep disorders screening. By conducting a collaborative study involving sleep medicine clinicians, sleep researchers, a consultant on alarms, together with the representatives from the management, and union leadership of the fire department, we expect we will develop a sleep optimization program with a high probability of success and test the hypotheses that increasing the sleep opportunity of firefighters will improve the alertness, performance, safety and physical and mental health of firefighters. The results of this study will provide policy makers with the scientific evidence they require to develop effective fatigue countermeasure programs for firefighters.

We will be conducting a randomized clinical trial, providing the most rigorous evaluation possible in an operational setting. Half the fire stations in a department will be randomly assigned to complete the intervention, termed Operation Fight Fatigue, in the first year of the study. The other half of the fire stations will complete the intervention in the second year. In this way, all firefighters will have the chance to benefit. We expect the fatigue countermeasure intervention to improve the alertness, performance, health and safety of firefighters. We will be evaluating a cost-effective intervention to improve the safety and health of firefighters in departments throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* Must be a fire department employee at a participating fire department.

Exclusion Criteria:

* May not be 17 years of age or younger.
* Will not be included if not a firefighter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Sleep and health screening of firefighters using a composite of survey instruments | The baseline survey will be conducted at the start of the study and the follow-up survey will be conducted approximately 12 months later.
  All firefighters in intervention and control stations will be asked to complete two surveys in which they document their work hours, sleep hours, sleep quality, caffeine consumption, and baseline health; their mood, sleepiness, and quality of life on a series of validated scales. Descriptions of any motor vehicle crashes, near miss crashes, and on-the-job injuries will also be obtained. Mental health will be assessed with three validated survey instruments. They will also receive the sleep disorders screening survey. Those found at high risk will be contacted to make aware.
Composite of firefighter information provided by the participating fire department | Up to 1 year
  The following outcomes will be collected: a) work hours data: scheduled work hours, overtime and vacation time; b) health and safety data: driving accidents and vehicle damage (including severity of accidents in terms of financial cost, time away from work, and extent of injury), on-the-job injuries (related and unrelated to motor vehicle crashes), sick time; and c) job performance data: response time and clear time (i.e., time to initial response and completion of a self-initiated or assigned task) and other measures considered pertinent to firefighters' performance by the department.
Sleep and performance of firefighters measured by a composite of physiological monitoring | Participants will be involved for up to 3 weeks and will have a follow-up physical exam (including blood work) up to 1 year later.
  Participants will participate in physiological monitoring to obtain objective data on sleep and performance. These data may also be used to validate the data reported on the survey. These firefighters will complete daily sleep/work diaries, wear an actigraph continuously and wear the Optalert glasses on the commute from each work shift. Subjects will also have 2 physical exams which include blood work.

SECONDARY OUTCOMES:
Documentation of motor vehicle crashes (MVC), and reported injuries | Up to 1 year
  If a participant reports a motor vehicle crash, or an occupational injury, he or she will be asked to describe the incident in detail, and provide copies of police records, automobile repair receipts, or insurance records for documentation.
Employment verification as a firefighter of all participants | Up to 1 year
  For the purposes of validating the study cohort approximately 10% may be randomly chosen to have their place of employment verified to ensure they are fire department employees. To do this our research staff will call, email, and/or send letters to the subject's place of employment asking to verify the status of the participant as either a past or present employee.
Composite of firefighter health information | Up to 1 year
  First, we request access to the accident and injury reports from the department-wide measures to look at overall changes in health and safety between the groups. Second, we will ask subjects to provide a written medical release to allow the researchers to gain access to the work physicals. Third, if a subject is found to be at high risk for a sleep disorder and takes a sleep clinic referral, we will ask them to provide a written medical release to allow access to their sleep clinic information. Fourth, we would request access to occupational health records.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Czeisler, PH.D., M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Division of Sleep Medicine; Brigham and Women's Hospital, Boston, Massachusetts, United States